CLINICAL TRIAL: NCT02302274
Title: Diagnostic Value and Safety of Flecainide Infusion Test in Brugada Syndrome
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 10-00253
Record Dates: First submitted 2014-11-24; First posted 2014-11-26 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Brugada Syndrome; Arrhythmogenic Right Ventricular Cardiomyopathy
Keywords: Brugada Syndrome; ARVC; flecainide; ST elevation
MeSH Terms: conditions — Brugada Syndrome; Arrhythmogenic Right Ventricular Dysplasia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- flecainide infusion test: Patients with suspect Brugada Syndrome will be asked to undergo flecainide infusion (2 mg/Kg up to 150 mg maximum dose) over 10 minutes and their ECG will be continuously monitored. The objective of the study is to investigate if they show conversion from type 2 or type 3 ECG to a diagnostic type 1 ECG.
  Interventions: Drug: flecainide iv

INTERVENTIONS:
Drug: flecainide iv — infusion over 10 min

SUMMARY:
The study aims to use flecainide infusion test as diagnostic test to unmask concealed Brugada Syndrome cases. It proposes to assess the safety profile of this test in US patients and its higher sensitivity when compared to procainamide infusion (the conventional drug used in the USA). As a substudy it proposes to apply this test to early ARVC cases in order to evaluate if ECG changes similar to those seen in Brugada Syndrome could be unmasked by flecainide iv.

DETAILED DESCRIPTION:
Brugada Syndrome is an inherited arrhythmogenic disease responsible for life-threatening arrhythmias and sudden cardiac death in young individuals with structural normal heart.

It is characterized by a peculiar ECG pattern, but this pattern could be intermittent. The infusion of sodium channel blockers (flecainide, ajmaline, procainamide) is used to unmask a concealed ECG pattern, thus providing an essential contribution to the diagnosis of this condition.

In the current clinical practice in USA, only procainamide is used for diagnostic purposes; however in Europe only ajmaline and flecainide, available as iv formulations, are widely used. European and Japanese studies have demonstrated that the use of flecainide harbors less risks of adverse events in patients and may have a higher accuracy in unraveling the presence of the disease.

In the present study the investigators propose to use flecainide infusion test in the Cardiovascular Genetics Program at NYUMC, in order to assess its sensitivity and specificity in diagnosing the disease and compare the incidence of adverse events to that observed during procainamide use.

Additionally, the investigators propose to extend the study protocol to patients with a suspect diagnosis of Arrhythmogenic Right Ventricular Tachycardia (ARVC), due to the possible overlap between the two conditions.

The study has the following aims:

1. To demonstrate the higher sensitivity and specificity of flecainide iv infusion compared to procainamide infusion for the diagnosis of Brugada Syndrome.
2. To demonstrate that flecainide is equally safe or safer than procainamide to use for diagnosing Brugada Syndrome.
3. To demonstrate that flecainide has high sensitivity and specificity in diagnosing also some patients with early stage Arrhythmogenic Right Ventricular Cardiomyopathy (ARVC).

ELIGIBILITY:
Inclusion Criteria:

* Suspect diagnosis of Brugada Syndrome or ARVC
* Idiopathic ventricular fibrillation and suspect concealed Brugada syndrome
* Family history of Brugada Syndrome
* Family history of unexpected cardiac sudden death

Exclusion Criteria:

* Type 1 Brugada Syndrome ECG
* Pregnancy
* History and/or evidence of ischemic cardiomyopathy
* Recent myocardial infarction
* Allergy or known adverse reaction to flecainide

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients (age>18) who are seen in the Cardiovascular Genetics Program with a suspect diagnosis of Brugada Syndrome or with a suspect diagnosis of ARVC. This study will enroll adult individuals who are referred to the Center with a suspect of Brugada Syndrome or ARVC on the basis of uncertain ECG pattern, family history for sudden death syncope and/or cardiac arrest and/or ventricular arrhythmia in the absence of clear clinical markers for any other inherited cardiac disease.
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2010-07-01; Primary Completion 2017-07-26 (Actual); Study Completion 2017-07-26 (Actual)

PRIMARY OUTCOMES:
diagnosis | 10 minutes
  conversion from type 2/3 Brugada ECG to diagnostic type 1 ECG

SECONDARY OUTCOMES:
absence of arrhythmias elicited during the test | 10 minutes
  number of arrhythmias caused by

CONTACTS AND LOCATIONS:
Overall Officials: Steven Fowler, MD, Principal Investigator — NYU School of Medicine
Locations (1):
- New york University, School of Medicine, New York, New York, United States